CLINICAL TRIAL: NCT05916586
Title: Effect of Short-Term Prednisone Therapy on C-reactive Protein Change in Emergency Department Patients With Acute Heart Failure and Elevated Inflammatory Markers
Brief Title: Effect of Short-term Prednisone Therapy on C-reactive Protein in Patients With Acute Heart Failure
Acronym: CORTAHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHF202301
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Heart Failure
Keywords: Acute Heart Failure; C-Reactive protein; Inflammation; Prednisone
MeSH Terms: conditions — Inflammation | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Parallel-group, comparative, open-label, randomised, controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone + usual care (Experimental): Prednisone tablets, 40 mg once a day orally, for 7 days plus usual treatment for acute heart failure
  Interventions: Drug: Prednisone
- Usual care (No Intervention): Usual treatment for acute heart failure

INTERVENTIONS:
Drug: Prednisone — Prednisone 40 mg orally once a day for 7 days
  Arms: Prednisone + usual care

SUMMARY:
This is a multicenter, parallel-group, randomized, open-label, controlled trial. Patients with a diagnosis of acute heart failure (AHF) in the emergency department (ED) or after emergency presentation to hospital will be screened and informed of the study. After signed consent, patients will be randomized into the control group (usual AHF treatment) or intervention group (usual AHF treatment + prednisone). Prednisone will be given for 7 days. Patients will be assessed at days 2, 4 or at discharge if earlier, and at day 7 at hospital visit. If the patient has been discharged before day 7, a follow-up visit will be scheduled at day 7 for endpoints assessment followed by a scheduled hospital visit at day 31 and a telephone follow-up at day 91. Study drug will be dispensed for the patient to take home until day 7.

DETAILED DESCRIPTION:
CORTAHF is a parallel-group, comparative, open-label, randomised (1:1), controlled trial. Patients with a diagnosis of AHF in the ED or after emergency presentation to hospital will be screened and informed of the study. After signed consent, patients will be randomized into the control group (usual AHF treatment) or intervention group (usual AHF treatment + prednisone).

Prednisone will be given for 7 days. Patients will be assessed at days 2, 4 or at discharge if earlier, and at day 7 at hospital visit. If the patient has been discharged before day 7, a follow-up visit will be scheduled at day 7 for endpoints assessment followed by a scheduled hospital visit at day 31 and a telephone follow-up at day 91. Study drug will be dispensed for the patient to take home until day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years of age
2. Unplanned ED visit or hospital presentation within the 12 hours prior to Screening with acute or worsening dyspnea and/or orthopnea, and pulmonary congestion on chest X-ray or lung ultrasound.
3. All measures from presentation to randomization of systolic blood pressure ≥ 100 mmHg, and of heart rate ≥ 60 bpm.
4. Written informed consent to participate in the study.
5. Biomarker levels indicative of congestion and inflammation: At Screening, NT-proBNP > 1,500 pg/mL and CRP > 20 mg/L
6. Patient agrees for follow-up visits at the hospital at day 7 in case of earlier discharge and Day 31.

Exclusion Criteria:

1. Anticipated life expectancy less than 6 months
2. Mechanical ventilation (not including CPAP/BIPAP) prior to Screening.
3. Significant pulmonary disease contributing substantially to the patients' dyspnea such as FEV1< 1 liter or need for chronic systemic or non-systemic steroid therapy, or any kind of primary right heart failure such as primary pulmonary hypertension or recurrent pulmonary embolism.
4. Myocardial infarction, unstable angina or cardiac surgery within 3 months, or cardiac resynchronization therapy (CRT) device implantation within 3 months, or percutaneous transluminal coronary intervention (PTCI), within 1 month prior to inclusion.
5. Index Event (admission for AHF) triggered primarily by a correctable etiology such as significant arrhythmia (e.g., sustained ventricular tachycardia, or atrial fibrillation/flutter with sustained ventricular response >130 beats per minute, or bradycardia with sustained ventricular arrhythmia <45 beats per minute), infection, severe anemia, acute coronary syndrome, pulmonary embolism, exacerbation of COPD, planned admission for device implantation or severe non-adherence leading to very significant fluid accumulation prior to admission and brisk diuresis after admission. Troponin elevations without other evidence of an acute coronary syndrome are not an exclusion.
6. Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
7. History of heart transplant or on a transplant list, or using or planned to be implanted with a ventricular assist device.
8. Sustained ventricular arrhythmia with syncopal episodes within the 3 months prior to screening that is untreated.
9. Presence at screening of any hemodynamically significant valvular stenosis or regurgitation, except mitral or tricuspid regurgitation secondary to left ventricular dilatation, or the presence of any hemodynamically significant obstructive lesion of the left ventricular outflow tract.
10. Primary liver disease considered to be life threatening
11. Renal disease or eGFR < 30 or > 80 mL/min/1.73m2 (as estimated by the simplified MDRD formula) at inclusion or history of dialysis.
12. Systemic steroid therapy, within 30 days from inclusion.
13. Inability to consent, or patient under guardianship measure
14. Participation in another intervention trial in the past 30 days
15. Anticipated non-adherence to study protocol or follow-up.
16. Pregnant or nursing (lactating) women.
17. Known hypersensitivity to steroids or constituents of prednisone tablets (excipients)
18. Psychotic states not yet controlled by treatment
19. Concomitant administration of live vaccines and up to 3 months after end of corticotherapy administration.
20. Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom
21. Persons subject to psychiatric care without their consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Change of CRP level | 7 days
  Change of CRP level, defined by CRP level at day 7 minus CRP level at inclusion.

SECONDARY OUTCOMES:
WHF adverse event, death, or hospital readmission | 91 days
  Time to first event of WHF adverse event, death, or hospital readmission for decompensated HF to day 91.
Change in quality of life | 7 days
  Changes in quality of life measured by the EQ-5D-5L from randomization to day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, MD, Principal Investigator — Emergency Department, Hôpital Universitaire Pitié-Salpêtrière, AP-HP, Paris, France
Locations (3):
- Armenia (3):
  - "Armenia" Republican Medical Center, Yerevan
  - "Mikaelyan" Surgery Institute, Yerevan
  - Erebouni Medical Center, Yerevan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrigo M, Jessup M, Mullens W, Reza N, Shah AM, Sliwa K, Mebazaa A. Acute heart failure. Nat Rev Dis Primers. 2020 Mar 5;6(1):16. doi: 10.1038/s41572-020-0151-7. PMID 32139695
- [Background] Burstin H. "Crossing the Quality Chasm" in emergency medicine. Acad Emerg Med. 2002 Nov;9(11):1074-7. doi: 10.1111/j.1553-2712.2002.tb01560.x. No abstract available. PMID 12414454
- [Background] Cannon JA, McKean AR, Jhund PS, McMurray JJ. What can we learn from RELAX-AHF compared to previous AHF trials and what does the future hold? Open Heart. 2015 Dec 23;2(1):e000283. doi: 10.1136/openhrt-2015-000283. eCollection 2015. PMID 26719808
- [Background] Cotter G, Dittrich HC, Weatherley BD, Bloomfield DM, O'Connor CM, Metra M, Massie BM; Protect Steering Committee, Investigators, and Coordinators. The PROTECT pilot study: a randomized, placebo-controlled, dose-finding study of the adenosine A1 receptor antagonist rolofylline in patients with acute heart failure and renal impairment. J Card Fail. 2008 Oct;14(8):631-40. doi: 10.1016/j.cardfail.2008.08.010. Epub 2008 Sep 14. PMID 18926433
- [Background] Davison BA, Senger S, Sama IE, Koch GG, Mebazaa A, Dickstein K, Samani NJ, Metra M, Anker SD, Cleland JG, Ng LL, Mordi IR, Zannad F, Filippatos GS, Hillege HL, Ponikowski P, van Veldhuisen DJ, Lang CC, van der Meer P, Nunez J, Bayes-Genis A, Edwards C, Voors AA, Cotter G. Is acute heart failure a distinctive disorder? An analysis from BIOSTAT-CHF. Eur J Heart Fail. 2021 Jan;23(1):43-57. doi: 10.1002/ejhf.2077. Epub 2021 Jan 22. PMID 33340221
- [Background] Du Clos TW. Function of C-reactive protein. Ann Med. 2000 May;32(4):274-8. doi: 10.3109/07853890009011772. PMID 10852144
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Freund Y, Cachanado M, Delannoy Q, Laribi S, Yordanov Y, Gorlicki J, Chouihed T, Feral-Pierssens AL, Truchot J, Desmettre T, Occelli C, Bobbia X, Khellaf M, Ganansia O, Bokobza J, Balen F, Beaune S, Bloom B, Simon T, Mebazaa A. Effect of an Emergency Department Care Bundle on 30-Day Hospital Discharge and Survival Among Elderly Patients With Acute Heart Failure: The ELISABETH Randomized Clinical Trial. JAMA. 2020 Nov 17;324(19):1948-1956. doi: 10.1001/jama.2020.19378. PMID 33201202
- [Background] Goonewardena SN, Stein AB, Tsuchida RE, Rattan R, Shah D, Hummel SL. Monocyte Subsets and Inflammatory Cytokines in Acute Decompensated Heart Failure. J Card Fail. 2016 May;22(5):358-65. doi: 10.1016/j.cardfail.2015.12.014. Epub 2015 Dec 17. PMID 26705751
- [Background] Kalogeropoulos AP, Tang WH, Hsu A, Felker GM, Hernandez AF, Troughton RW, Voors AA, Anker SD, Metra M, McMurray JJ, Massie BM, Ezekowitz JA, Califf RM, O'Connor CM, Starling RC, Butler J. High-sensitivity C-reactive protein in acute heart failure: insights from the ASCEND-HF trial. J Card Fail. 2014 May;20(5):319-26. doi: 10.1016/j.cardfail.2014.02.002. Epub 2014 Feb 12. PMID 24530944
- [Background] Le Conte P, Terzi N, Mortamet G, Abroug F, Carteaux G, Charasse C, Chauvin A, Combes X, Dauger S, Demoule A, Desmettre T, Ehrmann S, Gaillard-Le Roux B, Hamel V, Jung B, Kepka S, L'Her E, Martinez M, Milesi C, Morawiec E, Oberlin M, Plaisance P, Pouyau R, Raherison C, Ray P, Schmidt M, Thille AW, Truchot J, Valdenaire G, Vaux J, Viglino D, Voiriot G, Vrignaud B, Jean S, Mariotte E, Claret PG. Management of severe asthma exacerbation: guidelines from the Societe Francaise de Medecine d'Urgence, the Societe de Reanimation de Langue Francaise and the French Group for Pediatric Intensive Care and Emergencies. Ann Intensive Care. 2019 Oct 10;9(1):115. doi: 10.1186/s13613-019-0584-x. PMID 31602529
- [Background] Liu C, Liu G, Zhou C, Ji Z, Zhen Y, Liu K. Potent diuretic effects of prednisone in heart failure patients with refractory diuretic resistance. Can J Cardiol. 2007 Sep;23(11):865-8. doi: 10.1016/s0828-282x(07)70840-1. PMID 17876376
- [Background] Liu C, Ge N, Zhai JL, Zhang JX. Dexamethasone-induced diuresis is associated with inhibition of the renin-angiotensin-aldosterone system in rats. Kaohsiung J Med Sci. 2016 Dec;32(12):614-619. doi: 10.1016/j.kjms.2016.09.007. Epub 2016 Oct 27. PMID 27914612
- [Background] Liu C, Zhao Q, Zhen Y, Zhai J, Liu G, Zheng M, Ma G, Wang L, Tian L, Ji L, Li L, Duan L, Liu K. Effect of Corticosteroid on Renal Water and Sodium Excretion in Symptomatic Heart Failure: Prednisone for Renal Function Improvement Evaluation Study. J Cardiovasc Pharmacol. 2015 Sep;66(3):316-22. doi: 10.1097/FJC.0000000000000282. PMID 25992918
- [Background] Mebazaa A, Yilmaz MB, Levy P, Ponikowski P, Peacock WF, Laribi S, Ristic AD, Lambrinou E, Masip J, Riley JP, McDonagh T, Mueller C, deFilippi C, Harjola VP, Thiele H, Piepoli MF, Metra M, Maggioni A, McMurray J, Dickstein K, Damman K, Seferovic PM, Ruschitzka F, Leite-Moreira AF, Bellou A, Anker SD, Filippatos G. Recommendations on pre-hospital & early hospital management of acute heart failure: a consensus paper from the Heart Failure Association of the European Society of Cardiology, the European Society of Emergency Medicine and the Society of Academic Emergency Medicine. Eur J Heart Fail. 2015 Jun;17(6):544-58. doi: 10.1002/ejhf.289. Epub 2015 May 21. PMID 25999021
- [Background] Metra M, Teerlink JR, Cotter G, Davison BA, Felker GM, Filippatos G, Greenberg BH, Pang PS, Ponikowski P, Voors AA, Adams KF, Anker SD, Arias-Mendoza A, Avendano P, Bacal F, Bohm M, Bortman G, Cleland JGF, Cohen-Solal A, Crespo-Leiro MG, Dorobantu M, Echeverria LE, Ferrari R, Goland S, Goncalvesova E, Goudev A, Kober L, Lema-Osores J, Levy PD, McDonald K, Manga P, Merkely B, Mueller C, Pieske B, Silva-Cardoso J, Spinar J, Squire I, Stepinska J, Van Mieghem W, von Lewinski D, Wikstrom G, Yilmaz MB, Hagner N, Holbro T, Hua TA, Sabarwal SV, Severin T, Szecsody P, Gimpelewicz C; RELAX-AHF-2 Committees Investigators. Effects of Serelaxin in Patients with Acute Heart Failure. N Engl J Med. 2019 Aug 22;381(8):716-726. doi: 10.1056/NEJMoa1801291. PMID 31433919
- [Background] Nieminen MS, Dickstein K, Fonseca C, Serrano JM, Parissis J, Fedele F, Wikstrom G, Agostoni P, Atar S, Baholli L, Brito D, Colet JC, Edes I, Gomez Mesa JE, Gorjup V, Garza EH, Gonzalez Juanatey JR, Karanovic N, Karavidas A, Katsytadze I, Kivikko M, Matskeplishvili S, Merkely B, Morandi F, Novoa A, Oliva F, Ostadal P, Pereira-Barretto A, Pollesello P, Rudiger A, Schwinger RH, Wieser M, Yavelov I, Zymlinski R. The patient perspective: Quality of life in advanced heart failure with frequent hospitalisations. Int J Cardiol. 2015 Jul 15;191:256-64. doi: 10.1016/j.ijcard.2015.04.235. Epub 2015 May 1. PMID 25981363
- [Background] Oppe, M., R. Rabin, et al. (2008). EQ-5D User Guide. Version 1.0. Rotterdam, The Netherlands, The EuroQol Group.
- [Background] Raess N, Schuetz P, Cesana-Nigro N, Winzeler B, Urwyler SA, Schaedelin S, Rodondi N, Blum MR, Briel M, Mueller B, Christ-Crain M, Blum CA. Influence of Prednisone on Inflammatory Biomarkers in Community-Acquired Pneumonia: Secondary Analysis of a Randomized Trial. J Clin Pharmacol. 2021 Nov;61(11):1406-1414. doi: 10.1002/jcph.1914. Epub 2021 Jul 27. PMID 34031890
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Wedzicha JA Ers Co-Chair, Miravitlles M, Hurst JR, Calverley PM, Albert RK, Anzueto A, Criner GJ, Papi A, Rabe KF, Rigau D, Sliwinski P, Tonia T, Vestbo J, Wilson KC, Krishnan JA Ats Co-Chair. Management of COPD exacerbations: a European Respiratory Society/American Thoracic Society guideline. Eur Respir J. 2017 Mar 15;49(3):1600791. doi: 10.1183/13993003.00791-2016. Print 2017 Mar. PMID 28298398
- [Background] Yao TC, Huang YW, Chang SM, Tsai SY, Wu AC, Tsai HJ. Association Between Oral Corticosteroid Bursts and Severe Adverse Events : A Nationwide Population-Based Cohort Study. Ann Intern Med. 2020 Sep 1;173(5):325-330. doi: 10.7326/M20-0432. Epub 2020 Jul 7. PMID 32628532
- [Result] Biegus J, Cotter G, Davison BA, Freund Y, Voors AA, Edwards C, Novosadova M, Takagi K, Hayrapetyan H, Mshetsyan A, Mayranush D, Cohen-Solal A, Ter Maaten JM, Filippatos G, Chioncel O, Sadoune M, Pagnesi M, Simon T, Metra M, Mann DL, Mebazaa A, Ponikowski P. The Effects of Burst Steroid Therapy on Short-term Decongestion in Acute Heart Failure Patients With Pro-inflammatory Activation: A Post Hoc Analysis of the CORTAHF Randomized, Open-label, Pilot Trial. J Card Fail. 2025 Feb;31(2):354-366. doi: 10.1016/j.cardfail.2024.09.002. Epub 2024 Sep 29. PMID 39353506
- [Result] Pagnesi M, Cotter G, Davison BA, Freund Y, Voors AA, Edwards C, Novosadova M, Takagi K, Hayrapetyan H, Mshetsyan A, Drambyan M, Cohen-Solal A, Ter Maaten JM, Biegus J, Ponikowski P, Filippatos G, Chioncel O, Sadoune M, Simon T, Mann DL, Mebazaa A, Metra M. Burst steroid therapy and quality of life in patients with acute heart failure: Insights from the CORTAHF trial. ESC Heart Fail. 2025 Jun;12(3):1620-1629. doi: 10.1002/ehf2.15235. Epub 2025 Feb 11. PMID 39934967
- [Result] Cotter G, Davison B, Freund Y, Mebazaa A, Voors A, Edwards C, Novosadova M, Takagi K, Hayrapetyan H, Mshetsyan A, Mayranush D, Cohen-Solal A, Ter Maaten JM, Biegus J, Ponikowski P, Filippatos G, Chioncel O, Pagnesi M, Simon T, Metra M, Mann DL. Corticosteroid burst therapy in patients with acute heart failure: Design of the CORTAHF pilot study. ESC Heart Fail. 2024 Oct;11(5):2672-2680. doi: 10.1002/ehf2.14930. Epub 2024 Jun 28. PMID 38943232
- [Result] Cotter G, Davison BA, Freund Y, Voors AA, Edwards C, Novosadova M, Takagi K, Hayrapetyan H, Mshetsyan A, Mayranush D, Cohen-Solal A, Ter Maaten JM, Biegus J, Ponikowski P, Filippatos G, Chioncel O, Sadoune M, Pagnesi M, Simon T, Metra M, Mann DL, Mebazaa A. Burst steroid therapy for acute heart failure: The CORTAHF randomized, open-label, pilot trial. Eur J Heart Fail. 2024 Oct;26(10):2282-2292. doi: 10.1002/ejhf.3452. Epub 2024 Aug 30. PMID 39211989